CLINICAL TRIAL: NCT03981601
Title: the Histomorphometric Study of Nanocrystalline Hydroxyapatite (Nano Bone) With Lovastatin in the Preservation of the Tooth Socket
Brief Title: Evaluation, the Histomorphometric Study of Nanocrystalline Hydroxyapatite (Nano Bone) Wif Lovastatin in the Preservation of the Tooth Socket
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, assistant prof, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2038
Record Dates: First submitted 2019-02-09; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Lovastatin; Pharmaceutical Preparations; Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lovastatin 40 mg with bone graft (Active Comparator): after tooth extraction, put teh lovastatin40 mg wif bone graft wifin tooth socket
  Interventions: Drug: Lovastatin 40 MG
- without drug with bone graft (Active Comparator): after tooth extraction, put the bone graft wifin tooth socket
  Interventions: Procedure: without drug with Bone graft

INTERVENTIONS:
Drug: Lovastatin 40 MG — after tooth extraction, put teh lovastatin40 mg wif bone graft wifin tooth socket
  Other Names: Group A
  Arms: lovastatin 40 mg with bone graft
Procedure: without drug with Bone graft — after tooth extraction, put teh bone graft wifin tooth socket
  Other Names: Group B
  Arms: without drug with bone graft

SUMMARY:
Twenty patients referring to periodontics department of Boroujerd Azad university of dentistry after obtaining consent to participate in the research project, which have more than 20 teeth, are over 18 years old and require socket preservation surgery to tooth extraction for the periodontal problem, caries or Fractures were selected.

DETAILED DESCRIPTION:
twenty healthy patients referring to periodontics department of Boroujerd Azad university of dentistry after obtaining consent to participate in the research project, which has more than 20 teeth, are over 18 years old and require socket preservation surgery to tooth extraction for the periodontal problem, caries or Fractures were selected. moreover, divided the socket randomly to two groups(A, B)including A: bone graft with lovastatin and B: bone graft alone, after 3 months with trephine will collect the samples. following the histomorphometric analysis.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years old
2. tooth fracture, root caries
3. Patients are volunteered for placement of the implant

Exclusion Criteria:

1. systemic diseases
2. Pregnancy and breastfeeding
3. malignancy, radiation therapy,
4. history of periodontal surgery during the six months ago.
5. medicine(phosphonates, antibiotic,...)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Socket preservation with Lovastatin as evaluated by the amount of bone formation volume | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Amirhossein Farahmand, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No